CLINICAL TRIAL: NCT00083421
Title: Effects of ONO-2506PO in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-2506POU010
Record Dates: First submitted 2004-05-24; First posted 2004-06-18 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: ONO-2506PO

SUMMARY:
The purpose of this study is to establish the presence of an effect of treatment with ONO-2506PO in patients with Alzheimer's Disease, based upon cognitive and global scales.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's Disease using NINCDS/ADRDA criteria
* Standardized MMSE Score of 13 to 24 points (inclusive)
* Modified Hachinski score equal or less than 4

Exclusion Criteria:

* Serious systemic disease that may preclude survival to study completion
* Other illnesses that may include dementive features

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 647 (Actual)
Dates: Start 2004-06; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Cognitive Function Scale
Global Function Scale

SECONDARY OUTCOMES:
ADL Scale
Psychiatric Symptom Scale

CONTACTS AND LOCATIONS:
Locations (87):
- United States (79):
  - Kirkland Clinic, Birmingham, Alabama
  - Alzheimers Disease Research Center, Birmingham, Alabama
  - Pivotal Research Center, Mesa, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Sun Health Research Institute, Sun City, Arizona
  - University of Arizona, Tucson, Arizona
  - Margolin Brain Institute, Fresno, California
  - UCI Medical Center Neuropsychiatric Center, Orange, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - The Southwest Institute for Clinical Research, Inc, Rancho Mirage, California
  - Hamid Rabiee, MD, Redding, California
  - Alzheimers Disease Research Center, Univ of CA, San Diego, San Diego, California
  - Pacific Research Network, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Apex Research Institute, Santa Ana, California
  - Pacific Neuroscience Medical Group, Santa Barbara, California
  - Neurological Research Institute, Santa Monica, California
  - Radiant Research, Denver, Colorado
  - Research Center for Clinical Studies, Inc., Darien, Connecticut
  - GAP Clinical Care & Research Center, Hamden, Connecticut
  - Baumel-Eisner Neuromedical Institute, Boca Raton, Florida
  - Neurologic Consultants, Fort Lauderdale, Florida
  - Baumel-Eisner Neuromedical Institute, Fort Lauderdale, Florida
  - Gainsville Open MRI, Gainsville, Florida
  - Berma Research Group, Hialeah, Florida
  - Miami Jewish and Hospital for the Aged, Miami, Florida
  - Baumel-Eisner Neuromedical Institute, Miami Beach, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Research Site, Port Charlotte, Florida
  - Suncoast Neuroscience Associates, St. Petersburg, Florida
  - Meridien Research, St. Petersburg, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Johnnie B. Byrd Sr. Alzheimer's Center and Research Institute, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - DeKalb Neurology Associates, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Mercer University, Atlanta, Georgia
  - Rush Alzheimers Disease Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Radiant Research, Hoffman Estates, Illinois
  - Southern Illinois School of Medicine, Springfield, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Center for Alzheimers Disease and Related Disorders, Indianapolis, Indiana
  - Agewell, Indianapolis, Indiana
  - Louisiana State University Health Sciences Cntr - Dept of Psychiatry, New Orleans, Louisiana
  - J. Gary Booker, M.D., APMC, Shreveport, Louisiana
  - St. Louis University Medical Center, St Louis, Missouri
  - University of Nevada, Las Vegas, Nevada
  - Mid Atlantic Geriatric Association, Ocean Township, New Jersey
  - Meridian Institue for Aging, Paterson, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Upstate Clinical Reserach, LLC, Albany, New York
  - Upstate Neurology Consults, LLP, Albany, New York
  - Neurological Associates of Albany, Albany, New York
  - Neurobehavioral Research Inc., Lawrence, New York
  - Eastside Comprehensive Medical Services, New York, New York
  - Global Reserach & Consulting, Olean, New York
  - Monroe Community Hospital, Rochester, New York
  - Behavioral Medical Research, Staten Island, New York
  - Duke University Medical Center, Durham, North Carolina
  - Metrohealth Medical Center, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Infinity Research Group, LLC, Oklahoma City, Oklahoma
  - Clinical Pharmaceutical Trials, Tulsa, Oklahoma
  - Medford Neurological and Spine Clinic, Medford, Oregon
  - Summit Research Network, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Westmoreland Neurology Associates, Inc., Greensburg, Pennsylvania
  - University of PA, Section Geriatric Psychiatry, Philadelphia, Pennsylvania
  - Alzheimer Disease Research Center, Univ of Pittsburg, Pittsburgh, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Alzheimers Research and Clinical Programs, North Charleston, South Carolina
  - Claghorn Lesem Research Clinic, Bellaire, Texas
  - Memory Research Unit, Univ of Texas Southwest Med Ctr at Dallas, Dallas, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - Neurological Consultants, PC, Bennington, Vermont
  - Innovative Clinical Research Center, Alexandria, Virginia
  - Medical College of Wisconsin, Department of Neurology, Milwaukee, Wisconsin
  - Independent Psychiatric Consultants, Waukesha, Wisconsin
- Canada (8):
  - Inova Health Research, Inc., Kelowna, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia
  - Davidson Memory Clinic, Moncton, New Brunswick
  - Parkwood Hospital, Geriatric Medicine, London, Ontario
  - SCO Health Centre, Ottawa, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Pasqua Hospital, Regina, Saskatchewan